CLINICAL TRIAL: NCT00858637
Title: A Phase III, Multicentre, Double-blind, Double-dummy, Randomised, Flexible-dose, Comparative Study of MCI-196 Versus Simvastatin for the Treatment of Dyslipidaemia in Subjects With Chronic Kidney Disease on Dialysis (Incorporating a Placebo-controlled Withdrawal Phase)
Brief Title: Efficacy and Safety Study of MCI-196 Versus Simvastatin for Dyslipidaemia in Chronic Kidney Disease (CKD) Subjects on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-196-E11
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Dialysis; Dyslipidemia; Bile acid sequestrant
MeSH Terms: conditions — Renal Insufficiency, Chronic; Dyslipidemias | interventions — cholebine; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 MCI-196 (Experimental)
  Interventions: Drug: MCI-196; Drug: Placebo of Simvastatin
- 2 Placebo of MCI-196 (Placebo Comparator)
  Interventions: Drug: Placebo of Simvastatin; Drug: Placebo of MCI-196
- 3 Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin; Drug: Placebo of MCI-196
- 4 Placebo of Simvastatin (Placebo Comparator)
  Interventions: Drug: Placebo of Simvastatin; Drug: Placebo of MCI-196

INTERVENTIONS:
Drug: MCI-196 — Tablets of 3 g to 12 g/day (3 times a day) with dose escalation design during 16 weeks of Active Comparison Phase, and 4 weeks of fixed dose during Withdrawal Phase (Week 16 to Week 20)
  Other Names: Colestilan(INN); Colestimide(JAN); CHOLEBINE®; BindRen®
  Arms: 1 MCI-196
Drug: Placebo of Simvastatin — Tablets once a day, for 16 weeks of Active Comparison Phase, and 4 weeks of fixed dose during Withdrawal Phase (Week 16 to Week 20)
  Arms: 1 MCI-196; 2 Placebo of MCI-196; 4 Placebo of Simvastatin
Drug: Simvastatin — Tablets of 10 mg to 40 mg/day (once a day) with dose escalation design during 16 weeks of Active Comparison Phase, and 4 weeks of fixed dose during Withdrawal Phase (Week 16 to Week 20)
  Arms: 3 Simvastatin
Drug: Placebo of MCI-196 — Tablets 3 times a day for 16 weeks of Active Comparison Phase, and 4 weeks of fixed dose during Withdrawal Phase (Week 16 to Week 20)
  Arms: 2 Placebo of MCI-196; 3 Simvastatin; 4 Placebo of Simvastatin

SUMMARY:
The primary objective of this study is to demonstrate the superiority of MCI-196 over placebo and non-inferiority with simvastatin in reducing serum low-density lipoprotein (LDL)-cholesterol in subjects with chronic kidney disease Stage V on dialysis. This study incorporates a Washout Period and two treatment periods - an active comparison phase and a placebo-controlled withdrawal phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, and is >=18 years old
* Stable hemodialysis or peritoneal dialysis
* Subjects undergoing regular dialysis treatment
* If Female and of child-bearing potential, have a negative serum pregnancy test
* Male subjects must agree to use appropriate contraception

Exclusion Criteria:

* Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose him/her to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study
* Serum albumin level < 30 g/L
* Triglycerides level > 6.76 mmol/L (600 mg/dL)
* LDL-cholesterol level > 4.94 mmol/L (190 mg/dL)
* A History of significant gastrointestinal motility problems
* Biliary obstruction or proven liver dysfunction
* A positive test for HIV 1 and 2 antibodies
* A history of substance or alcohol abuse within the last year
* The subject has a history of rhabdomyolysis or myopathy
* Schedule to receive a kidney transplant within the next 6 months
* The subject has porphyria
* Participation in a clinical study with any experimental medication in the last 30 days or an experimental biological product within the last 90 days prior to signing of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (39):
- Belarus (5):
  - Brest
  - Grodno
  - Homyel
  - Minsk
  - Vitebsk
- Bulgaria (3):
  - Gabrovo
  - Plovdiv
  - Sofia
- Croatia (2):
  - Karlovac
  - Osijek
- Denmark (2):
  - Esbjerg
  - Roskilde
- Indonesia (5):
  - Jakarta
  - Malang
  - Medan
  - Palembang
  - Tamanlarea Makassar
- Israel (2):
  - Ashkelon
  - Nahariya
- Italy (6):
  - Bellano
  - Catania
  - Lecco
  - Merate
  - Milan
  - Oggiono
- Latvia (2):
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Kedauniai
  - Vilnius
- Malaysia (4):
  - George Town
  - Johor Bahru
  - Kelantan
  - Perak
- Romania (2):
  - Bucharest
  - Timișoara
- Singapore, Singapore
- Thailand (2):
  - Bangkok
  - Phitsanulok

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase: Active Comparison Phase: 3, 6, 9, 12g of MCI-196 / day as titrated
  * There was a gap of 1 subject between "STARTED" and "Overall Number of Baseline Participants".
  * One subject (A) was randomised to simvastatin (active) group but was dispensed MCI-196 in error at Week 12. This subject was counted as "STARTED" of Simvastatin (Active) group but counted as "Baseline Participants" of MCI-196 (active) group.
- MCI-196 (Active) + Simvastin (Placebo)/ Withdrawal Phase; MCI-196 (Placebo) + Simvastin (Placebo)/ Withdrawal Phase; Simvastin (Active) + MCI-196 (Placebo)/ Withdrawal Phase; Simvastin (Placebo) + MCI-196 (Placebo)/ Withdrawal Phase: Placebo-controlled Withdrawal Phase: dose level at the end of dose titration in the flexible dose period
- Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase: Active Comparison Phase: 10 mg to 40 mg of Simvastatin / day as titrated
  * There was a gap of 2 subject between "STARTED" and "Overall Number of Baseline Participants".
  * One subject did not take any study medication and excluded from "Baseline Participants".
  * In addition, one subject (A) was randomised to simvastatin (active) group but was dispensed MCI-196 in error at Week 12. This subject was counted as "STARTED" of Simvastatin (Active) group but counted as "Baseline Participants" of MCI-196 (active) group.
Period: Active Comparison Phase
Arm/Group | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase | MCI-196 (Active) + Simvastin (Placebo)/ Withdrawal Phase | MCI-196 (Placebo) + Simvastin (Placebo)/ Withdrawal Phase | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase | Simvastin (Active) + MCI-196 (Placebo)/ Withdrawal Phase | Simvastin (Placebo) + MCI-196 (Placebo)/ Withdrawal Phase
Started | 127 | 0 | 0 | 133 | 0 | 0
Completed | 103 | 0 | 0 | 115 | 0 | 0
Not Completed | 24 | 0 | 0 | 18 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0 | 9 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 6 | 0 | 0
Not completed — Other Reasons | 1 | 0 | 0 | 1 | 0 | 0
Period: Placebo-controlled Withdrawal Phase
Arm/Group | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase | MCI-196 (Active) + Simvastin (Placebo)/ Withdrawal Phase | MCI-196 (Placebo) + Simvastin (Placebo)/ Withdrawal Phase | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase | Simvastin (Active) + MCI-196 (Placebo)/ Withdrawal Phase | Simvastin (Placebo) + MCI-196 (Placebo)/ Withdrawal Phase
Started | 0 | 49 | 54 | 0 | 56 | 59
Completed | 0 | 49 | 53 | 0 | 55 | 58
Not Completed | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase | Total
Number analyzed (Participants) | 128 | 131 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (14.1) | 54.2 (13.6) | 53.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 61 | 120
  Male | 69 | 70 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum LDL-cholesterol Levels From Week 16 to Week 20 (LOCF) (ITT2)
Description: Percent Change from Week 16 to Week 20 (LOCF)
Time Frame: week20 minus week16
Population: ITT2 population included all re-randomised subjects who completed 16 weeks in the active treatment groups (MCI-196 or simvastatin), received at least 1 dose of study medication in the Placebo-controlled withdrawal phase and had at least 1 central serum LDL-C value after Week 16.
Measure: Mean (Standard Deviation); unit: Percent Change of LDL-cholesterol
Arm/Group | MCI-196 (Active) + Simvastin (Placebo)/ Withdrawal Phase | MCI-196 (Placebo) + Simvastin (Placebo)/ Withdrawal Phase | Simvastin (Active) + MCI-196 (Placebo)/ Withdrawal Phase | Simvastin (Placebo) + MCI-196 (Placebo)/ Withdrawal Phase
Number analyzed (Participants) | 49 | 53 | 55 | 58
Percent Change of LDL-cholesterol | 4.03 (19.92) | 42.55 (30.96) | 2.76 (18.43) | 49.84 (41.89)

2. Secondary Outcome: Percent Change in Serum LDL-cholesterol Levels From Baseline to Week 16 (LOCF) (ITT1)
Description: Percent Change from Baseline to Week 16 (LOCF)
Time Frame: week16 minus week0
Population: ITT1 population included all subjects who received a randomisation number, took at least 1 dose of study medication and had at least 1 central serum LDL-C value after the start of study medication.
Measure: Mean (Standard Deviation); unit: Percent Change of LDL-cholesterol
Groups:
- MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase: Active Comparison Phase: 3, 6, 9, 12g of MCI-196 / day as titrated
- Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase: Active Comparison Phase: 10 mg to 40 mgof Simvastatin / day as titrated
Arm/Group | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase
Number analyzed (Participants) | 125 | 127
Percent Change of LDL-cholesterol | -25.67 (19.45) | -26.38 (22.9)

3. Secondary Outcome: Change in Phosphorus(P), Calcium(Ca), Calcium-phosphorus Ion Product(PxCa) and Parathyroid Hormone (PTH)
Time Frame: 16 weeks and 20 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Vital Signs, Adverse Events, and Laboratory Values
Time Frame: throughout study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 16 weeks (Baseline - 16 weeks)
Description: Baseline Characteristics are reported based on the safety population, which is the actual number of participants that received each intervention. Details are described in [Arm/Group Description] of [Baseline Characteristics]
Groups:
- Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase: Active Comparison Phase: 10 mg to 40 mg of Simvastatin / day as titrated
Arm/Group | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase
Serious Adverse Events (participants affected / at risk) | 16/128 | 12/131
Other Adverse Events (participants affected / at risk) | 89/128 | 87/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase (N=128) | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase (N=131)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (Active) + Simvastatin (Placebo)/ Comparison Phase (N=128) | Simvastatin (Active) + MCI-196 (Placebo)/ Comparion Phase (N=131)
Anaemia (Blood and lymphatic system disorders) | 11 | 12
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve calcification (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 5 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Aerophagia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 10 | 7
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastric disorder (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 2 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 12
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 1 | 1
Hyperthermia (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 4 | 2
Pyrexia (General disorders) | 0 | 3
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 2 | 7
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 5 | 5
Procedural hypotension (Injury, poisoning and procedural complications) | 5 | 8
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood parathyroid hormone increased (Investigations) | 1 | 1
Blood phosphorus increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Lipids increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 12 | 6
Paraesthesia (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tonic convulsion (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 6 | 8
Hypertensive crisis (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 10 | 9
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other